CLINICAL TRIAL: NCT00465712
Title: Effect of Amnioinfusion on External Cephalic Version After Initial Failure a Prospective Multicentric Randomized Study
Brief Title: Effect of Amnioinfusion on External Cephalic Version Successful Rate
Acronym: AMNIO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRN05-FP/AMNIO2006
Record Dates: First submitted 2007-04-24; First posted 2007-04-25 (Estimated); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Breech Presentation
Keywords: transabdominal amnioinfusion; external cephalic version; breech presentation
MeSH Terms: conditions — Breech Presentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Transabdominal amnioinfusion performed before external cephalic version
  Interventions: Procedure: transabdominal amnioinfusion
- V (No Intervention): Without transabdominal amnioinfusion

INTERVENTIONS:
Procedure: transabdominal amnioinfusion — transabdominal amnioinfusion performed 4 to 24 hours before the second trial of external cephalic version
  Arms: A

SUMMARY:
The aim of the study is to evaluate the effect of transabdominal amnioinfusion before second external cephalic version after initial failure.Patient with a single foetus, at term, in breech presentation and after a first cephalic version are included. The randomisation determines whether the patient is included in the group with amnioinfusion before second cephalic version or with usual second cephalic version only; The efficacy's evaluation is based on rate of cephalic presentation at birth.Success rate of cephalic version with or without transabdominal amnioinfusion, rates of cesarian section in the two groups,maternal and fetal morbidity, time between second cephalic version and birth will be studied.

Prospective interventional randomized sequential comparative multicentric study. A maximum of 240 patients will be included (120 in each group). As the study is sequential it will be over as soon as a significative difference is shown.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the effect of transabdominal amnioinfusion before a second external cephalic version after initial failure. In case of success it could be an alternative to cesarian section. Without any other technique the foetus is in cephalic presentation after a first external cephalic version in 50%.

Patients with a single fetus, at term, in breech presentation are proposed to participate. The randomization is done at the inclusion and determines whether the patient is included in the group with amnioinfusion before second cephalic version or usual second cephalic version only. The only difference between the two groups is the realisation of an amnioinfusion, the cephalic version's technique is the same.

Efficacy's evaluation is based on rate of cephalic presentation at birth. Success rate of cephalic version, rates of cesarian section, maternal and fetal morbidity in the two groups, time between second cephalic version and birth will be studied.

ELIGIBILITY:
Inclusion Criteria:

* single fetal pregnancy
* breech presentation
* at term
* initial failure of external cephalic version
* structurally normal foetus

Exclusion Criteria:

* polyhydramnios
* anhydramnios
* abnormality of the fetal heart rhythm
* uterine congenital malformation
* cesarian section for a previous birth
* unability to understand study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2006-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
cephalic presentation at birth | at birth

CONTACTS AND LOCATIONS:
Overall Officials: Franck Perrotin, MD-PhD, Principal Investigator — Tours University Hospital
Locations (2):
- France (2):
  - Mother Child University Hospital, Nantes
  - Olympe de Gouges Women Health Centre, Bretonneau University Hospital, Tours

REFERENCES:
- [Background] Benifla JL, Goffinet F, Darai E, Madelenat P. Antepartum transabdominal amnioinfusion to facilitate external cephalic version after initial failure. Obstet Gynecol. 1994 Dec;84(6):1041-2. PMID 7970462
- [Background] Benifla JL, Goffinet F, Bascou V, Darai E, Proust A, Madelenat P. [Transabdominal amnio-infusion facilitates external version maneuver after initial failure. Six successful attempts]. J Gynecol Obstet Biol Reprod (Paris). 1995;24(3):319-22. French. PMID 7622781
- [Background] Boucher M, Bujold E, Marquette GP, Vezina Y. The relationship between amniotic fluid index and successful external cephalic version: a 14-year experience. Am J Obstet Gynecol. 2003 Sep;189(3):751-4. doi: 10.1067/s0002-9378(03)00846-9. PMID 14526307
- [Background] Cheng M, Hannah M. Breech delivery at term: a critical review of the literature. Obstet Gynecol. 1993 Oct;82(4 Pt 1):605-18. PMID 8377990
- [Background] Collaris RJ, Oei SG. External cephalic version: a safe procedure? A systematic review of version-related risks. Acta Obstet Gynecol Scand. 2004 Jun;83(6):511-8. doi: 10.1111/j.0001-6349.2004.00347.x. PMID 15144330
- [Background] Collea JV, Chein C, Quilligan EJ. The randomized management of term frank breech presentation: a study of 208 cases. Am J Obstet Gynecol. 1980 May 15;137(2):235-44. doi: 10.1016/0002-9378(80)90780-2. PMID 7377243
- [Background] Fernandez CO, Bloom SL, Smulian JC, Ananth CV, Wendel GD Jr. A randomized placebo-controlled evaluation of terbutaline for external cephalic version. Obstet Gynecol. 1997 Nov;90(5):775-9. doi: 10.1016/S0029-7844(97)00440-7. PMID 9351763
- [Background] Fischer R. Breech Presentation. 2004. http://www.emedicine.com/med/topic3272.htm
- [Background] Fisk NM, Ronderos-Dumit D, Soliani A, Nicolini U, Vaughan J, Rodeck CH. Diagnostic and therapeutic transabdominal amnioinfusion in oligohydramnios. Obstet Gynecol. 1991 Aug;78(2):270-8. PMID 2067774
- [Background] Flamm BL, Fried MW, Lonky NM, Giles WS. External cephalic version after previous cesarean section. Am J Obstet Gynecol. 1991 Aug;165(2):370-2. doi: 10.1016/0002-9378(91)90095-9. PMID 1872341
- [Background] Gembruch U, Hansmann M. Artificial instillation of amniotic fluid as a new technique for the diagnostic evaluation of cases of oligohydramnios. Prenat Diagn. 1988 Jan;8(1):33-45. doi: 10.1002/pd.1970080105. PMID 3278306
- [Background] Gimovsky ML, Wallace RL, Schifrin BS, Paul RH. Randomized management of the nonfrank breech presentation at term: a preliminary report. Am J Obstet Gynecol. 1983 May 1;146(1):34-40. doi: 10.1016/0002-9378(83)90923-7. PMID 6342396
- [Background] Gramellini D, Fieni S, Kaihura C, Faiola S, Vadora E. Transabdominal antepartum amnioinfusion. Int J Gynaecol Obstet. 2003 Nov;83(2):171-8. doi: 10.1016/s0020-7292(03)00274-1. PMID 14550592
- [Background] Gramellini D, Fieni S, Kaihura C, Piantelli G, Verrotti C. Antepartum amnioinfusion: a review. J Matern Fetal Neonatal Med. 2003 Nov;14(5):291-6. doi: 10.1080/jmf.14.5.291.296. PMID 14986801
- [Background] Gramellini D, Fieni S, Piantelli G, Faiola S, Kaihura C, Verrotti C, Cavallotti D, Viola P, Bacchini G, Vadora E. [Amnioinfusion: techniques, indications, and controlled retrospective study of 55 cases]. Acta Biomed Ateneo Parmense. 2000;71 Suppl 1:325-9. Italian. PMID 11424764
- [Background] Hannah ME, Hannah WJ, Hewson SA, Hodnett ED, Saigal S, Willan AR. Planned caesarean section versus planned vaginal birth for breech presentation at term: a randomised multicentre trial. Term Breech Trial Collaborative Group. Lancet. 2000 Oct 21;356(9239):1375-83. doi: 10.1016/s0140-6736(00)02840-3. PMID 11052579
- [Background] Hellstrom AC, Nilsson B, Stange L, Nylund L. When does external cephalic version succeed? Acta Obstet Gynecol Scand. 1990;69(4):281-5. doi: 10.3109/00016349009036147. PMID 2244457
- [Background] Hofmeyr GJ. Interventions to help external cephalic version for breech presentation at term. Cochrane Database Syst Rev. 2004;(1):CD000184. doi: 10.1002/14651858.CD000184.pub2. PMID 14973948
- [Background] Hofmeyr GJ, Hannah ME. Planned caesarean section for term breech delivery (Cochrane Review). In: The Cochrane Library, Issue 3, 2004b. Chichester, UK: John Wiley & Sons, Ltd
- [Background] Hofmeyr GJ, Kulier R. Cephalic version by postural management for breech presentation. Cochrane Database Syst Rev. 2000;(3):CD000051. doi: 10.1002/14651858.CD000051. PMID 10908458
- [Background] Hofmeyr GJ, Kulier R. External cephalic version for breech presentation at term (Cochrane Review). In: The Cochrane Library, Issue 3, 2004d. Chichester, UK: John Wiley & Sons, Ltd
- [Background] Hofmeyr GJ. External cephalic version facilitation for breech presentation at term. Cochrane Database Syst Rev. 2000;(2):CD000184. doi: 10.1002/14651858.CD000184. PMID 10796176
- [Background] Hofmeyr GJ. External cephalic version for breech presentation before term (Cochrane Review). In: The Cochrane Library, Issue 3, 2004e. Chichester, UK: John Wiley & Sons, Ltd.
- [Background] Hutton EK, Kaufman K, Hodnett E, Amankwah K, Hewson SA, McKay D, Szalai JP, Hannah ME. External cephalic version beginning at 34 weeks' gestation versus 37 weeks' gestation: a randomized multicenter trial. Am J Obstet Gynecol. 2003 Jul;189(1):245-54. doi: 10.1067/mob.2003.442. PMID 12861170
- [Background] Kotaska A. Inappropriate use of randomised trials to evaluate complex phenomena: case study of vaginal breech delivery. BMJ. 2004 Oct 30;329(7473):1039-42. doi: 10.1136/bmj.329.7473.1039. PMID 15514356
- [Background] Lansac J, Body G, Perrotin F, Marret H. Pratique de l'accouchement. Paris: Masson ; 2001, p. 365-369.
- [Background] Le Bret T, Grange G, Goffinet F, Cabrol D. [External cephalic version: experience about 237 versions at Port-Royal maternity]. J Gynecol Obstet Biol Reprod (Paris). 2004 Jun;33(4):297-303. doi: 10.1016/s0368-2315(04)96458-7. French. PMID 15170425
- [Background] Lilford RJ, van Coeverden de Groot HA, Moore PJ, Bingham P. The relative risks of caesarean section (intrapartum and elective) and vaginal delivery: a detailed analysis to exclude the effects of medical disorders and other acute pre-existing physiological disturbances. Br J Obstet Gynaecol. 1990 Oct;97(10):883-92. doi: 10.1111/j.1471-0528.1990.tb02442.x. PMID 2223678
- [Background] Newman RB, Peacock BS, VanDorsten JP, Hunt HH. Predicting success of external cephalic version. Am J Obstet Gynecol. 1993 Aug;169(2 Pt 1):245-9; discussion 249-50. doi: 10.1016/0002-9378(93)90071-p. PMID 8362933
- [Background] Novakov-Mikic A, Stojic S, Bogavac M, Mandic A. [Amnionic infusion therapy in conditions with low amnionic fluid levels]. Med Pregl. 2003 Jan-Feb;56(1-2):33-7. doi: 10.2298/mpns0302033n. Croatian. PMID 12793184
- [Background] Perrotin F, Sauget S, Laffont M, Lansac J, Body G. Version par manœuvre externe: nouveaux apports techniques. In: Collège National des Gynécologues Obstétriciens Français. Mises à jour en Gynécologie Obstétrique - VIGOT Ed. - Paris, 2003;25:5-23
- [Background] Pritchard JA, MacDonald PC. Dystocia caused by abnormalities in presentation, position, or development of the fetus. Williams Obstetrics. Norwalk, CT: Appleton-Century-Crofts; 1980, p. 787-796.
- [Background] Rietberg CC, Elferink-Stinkens PM, Brand R, van Loon AJ, Van Hemel OJ, Visser GH. Term breech presentation in The Netherlands from 1995 to 1999: mortality and morbidity in relation to the mode of delivery of 33824 infants. BJOG. 2003 Jun;110(6):604-9. PMID 12798480
- [Background] Royal College of Obstetricians and Gynaecologists Clinical Audit Unit. Effective procedures in maternity care suitable for audit. London: RCOG Press; 1997;4(7). Breech presentation at term, p. 32.
- [Background] Royal College of Obstetricians and Gynaecologists The management of breech presentation. 2001
- [Background] Royal College of Obstetricians and Gynaecologists. Use of anti-D immunoglobulin for Rh Prophylaxis. London: RCOG Press; 1999. Guideline n° 22
- [Background] Shalev E, Battino S, Giladi Y, Edelstein S. External cephalic version at term--using tocolysis. Acta Obstet Gynecol Scand. 1993 Aug;72(6):455-7. doi: 10.3109/00016349309021134. PMID 8394624
- [Background] Stuart IP. Term breech trial. Lancet. 2001 Jan 20;357(9251):228. doi: 10.1016/S0140-6736(05)71325-8. No abstract available. PMID 11213120
- [Background] Wagner A, Potin J, Himily V, Arbeille P, Perrotin F. The "Loss Of Resistance" Syringe: a useful tool for difficult amnioinfusion. Fetal Diagn Ther (submitted).
- [Background] Mousa HA. Re: Ledee et al. Management in intractable obstetric haemorrhage: an audit study on 61 cases. Eur J Obstet Gynecol Reprod Biol 2001;94:189-96. Eur J Obstet Gynecol Reprod Biol. 2001 Dec 10;100(1):116-7. doi: 10.1016/s0301-2115(01)00438-9. No abstract available. PMID 11728673
- [Background] Zhang J, Bowes WA Jr, Fortney JA. Efficacy of external cephalic version: a review. Obstet Gynecol. 1993 Aug;82(2):306-12. PMID 8336883
- [Result] Diguisto C, Winer N, Descriaud C, Tavernier E, Weymuller V, Giraudeau B, Perrotin F. Amnioinfusion for women with a singleton breech presentation and a previous failed external cephalic version: a randomized controlled trial. J Matern Fetal Neonatal Med. 2018 Apr;31(8):993-999. doi: 10.1080/14767058.2017.1304909. Epub 2017 Mar 28. PMID 28279119